CLINICAL TRIAL: NCT06379529
Title: The COPD CARE Study: Evaluating the Impact of a Virtual-First COPD Service on Major Cardiac and Respiratory Events
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuvoAir Medical PC (Industry)
Collaborators: Optum, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USCOPD2022B
Record Dates: First submitted 2023-08-25; First posted 2024-04-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: COPD Exacerbation; COPD; Cardio/Pulm: Heart Failure
Keywords: COPD; COPD Exacerbation; COPD Hospitalization; COPD Readmission; COPD Costs; Medicare; Medicare Advantage
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Pragmatic evaluation of a clinical service using a prospective cohort comparison of intervention vs propensity matched controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NuvoAir clinical service (Experimental): Patients with COPD receiving usual care plus the NuvoAir clinical service.The NuvoAir clinical service offers comprehensive remote monitoring of health parameters and patient-reported outcomes as well as personalized clinical and behavioral interventions tailored to the patients' unique needs and clinical risk. The service involves virtual interaction with NuvoAir coaches who provide guidance and assistance in navigating and utilizing the service; dedicated NuvoAir care coordinators for self-management support and educational resources, aiming to enhance the management of COPD and other comorbidities including cardiovascular conditions. In situations where patients encounter new or worsening symptoms, the NuvoAir clinical team is accessible to advise and triage as required.
  Interventions: Other: NuvoAir clinical service
- Standard Care (No Intervention): Propensity matched controls with COPD who receive usual care.

INTERVENTIONS:
Other: NuvoAir clinical service — Patients with COPD receiving usual care plus NuvoAir clinical services.
  Arms: NuvoAir clinical service

SUMMARY:
A 12 month interventional study of up to 1,050 people with COPD to determine if the NuvoAir virtual-first clinical service leads to fewer moderate and severe COPD exacerbations and cardiac events, reduces healthcare utilization, and lowers the total cost of care compared to a control cohort that receives standard care only.

DETAILED DESCRIPTION:
A virtual (decentralized), pragmatic, prospective, matched cohort study conducted in patients with COPD residing in the United States of America who are enrolled with one or more health insurers or providers supporting the study. The study aims to evaluate COPD outcomes with the addition of the NuvoAir virtual-first clinical service compared to a cohort receiving standard care (matched control - no intervention).

Each patient in the NuvoAir cohort will receive routine clinical care from their providers with the addition of the NuvoAir clinical service. The NuvoAir clinical service offers comprehensive monitoring of health parameters and patient-reported outcomes as well as personalized clinical and behavioral interventions tailored to the patients' unique needs and clinical risk. The service involves virtual interaction with NuvoAir coaches who provide guidance and assistance in navigating and utilizing the service. Dedicated NuvoAir care coordinators are available to offer self-management support and educational resources, aiming to enhance the management of COPD and comorbidities such as cardiovascular conditions. In situations where patients encounter new or worsening symptoms, the NuvoAir clinical team is accessible to provide advice and triage, as required.

Each patient in the standard care cohort will receive their routine clinical care from their healthcare provider. Only de-identified data that is usually collected by their health insurer or provider will be subject to analysis, no additional data will be collected for the standard care cohort.

NuvoAir and standard care cohorts will be matched on the basis of age, gender, disease severity (ICD10 code for COPD with a severe exacerbation of COPD in the previous 12 months or disease severity score of 2 or 3 as defined by their health plan) and period of entry into the study. Eligible patients will be recruited from Medicare patients in Medicare Advantage plans that are administered by the private health insurance company or health care provider supporting the study.

Key Objectives: To determine if use of the NuvoAir clinical service results in a reduction in the rate and number of moderate and severe exacerbations of COPD; major cardiac events; hospitalizations and 30-day readmissions; days hospitalized; and lowers healthcare costs compared with the matched cohort of patients receiving standard care only.

Study duration: The overall study duration is expected to be two years with one year of active patient participation using the NuvoAir clinical service following the end of the baseline period. This will be followed by one year of follow-up by reference to health insurer or provider's records.

Enrollment: The study will enroll up to 350 patients for the NuvoAir intervention and 700 for the standard care cohort for a total of 1,050 patients.

ELIGIBILITY:
Inclusion Criteria:

* Twelve months of claims data in the health insurer or provider's database for baseline
* ICD10 code for COPD (including emphysema and chronic bronchitis) with a severe exacerbation of COPD in the previous 12 months (defined as ER visit or hospitalization related to COPD or severity score of 2 or 3)
* Cooperative, i.e., subject should be able to follow and understand instructions
* Access to a phone (smartphone, cell phone, or landline)
* Willingness to sign a medical release form for treating healthcare facilities

Exclusion Criteria:

* Does not have access to a a phone (smartphone, cell phone, or landline)
* Lack of cooperation, subject cannot follow and understand instructions
* Other serious medical illness that, in the opinion of the PI, would interfere with the patient's participation in the study or interpretation of their data (i.e., terminal illness, unstable psychiatric condition, etc.)
* Does not understand English

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Moderate & Severe Exacerbations | 12 months
  Rate of moderate and severe exacerbations of COPD, measured by the health insurer or provider's records

SECONDARY OUTCOMES:
Severe COPD Exacerbations | 12 months
  Proportion of patients with at least one episode of severe COPD exacerbation within a 12-month period, NuvoAir cohort vs standard care cohort
Major Adverse Cardiac Event | 12 months
  Proportion of patients using the NuvoAir clinical service who have experienced a major adverse cardiac event (including CHF exacerbations, ACS/AMI, stroke) or all cause death, compared with the standard care cohort, measured using health insurer or provider records and assessed each year of the study
30-Day COPD Related Readmissions | 12 months
  Number of readmissions due to COPD exacerbation within a 30 day period following a COPD exacerbation (NuvoAir cohort only), compared to baseline and the number of 30-day readmissions after hospitalisation due to a COPD exacerbation compared to the standard care cohort
All-Cause Hospitalizations | 12 months
  Proportion of patients using the NuvoAir clinical service who have experienced an all-cause admission to hospital, compared with the standard care cohort, measured using health insurer or provider records and assessed each year of the study
All-Cause Readmissions | 12 months
  Number of all cause readmissions within a 30 day period following a COPD exacerbation, compared with the standard care cohort
Days Hospitalized due to COPD | 12 months
  Total number of days hospitalized due to COPD exacerbation, compared to the standard care cohort
Cost of Care Related to COPD | 12 months
  Cost of care related to COPD, including hospitalization, emergency room visits, urgent care visits, hospital visits, outpatient visits, and pharmacy costs, for those using NuvoAir Home compared with the standard care cohort
Medication Adherence | 12 months
  Percentage of the total doses of medication taken, which is the number of doses taken within a given time divided by the number of doses prescribed by a physician during the same time in NuvoAir cohort only
Quality of Life (QOL) | 12 months
  Quality of life measured using the SGRQ-C collected at baseline and at the end of the study

OTHER OUTCOMES:
Short-Acting Beta-Agonists Used | 12 months
  Number of short-acting beta-agonists used in one year from health insurer or provider records compared with the standard care cohort
Courses of Oral Antibiotics/Steroids | 12 months
  Number of courses of oral antibiotics/steroids in one year from health insurer or provider records compared with the standard care cohort
Self-efficacy | 12 months
  Self-efficacy for managing chronic disease scale score baseline vs end of study in NuvoAir cohort only
Patient Activation | 12 months
  Patient activation measure score baseline vs end of study in NuvoAir cohort only
Cat Score | 12 months
  CAT score baseline vs end of study in NuvoAir cohort only
mMRC Dyspnea Scale | 12 months
  mMRC dyspnea scale score baseline vs end of study in NuvoAir cohort only
Physical Activity | 12 months
  Average number of steps per day during the 2 week baseline period vs the average number of steps per day during a 2 week period 12 months later in NuvoAir cohort only

CONTACTS AND LOCATIONS:
Overall Officials: Ken Cohen, MD, Principal Investigator — Executive Director of Translational Research, OptumCare

IPD SHARING:
Plan to Share IPD: No